CLINICAL TRIAL: NCT04011891
Title: Comparison of OpeN VErsus RoboTic Partial Nephrectomy Trial - a Feasibility Randomized Controlled Trial
Brief Title: Comparison of OpeN VErsus RoboTic Partial Nephrectomy
Acronym: CONVERT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The Ontario government is now funding robotic partial nephrectomies.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18-5885
Record Dates: First submitted 2019-05-20; First posted 2019-07-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Renal Masses
Keywords: Minimally Invasive Surgery; Robotic Surgery; Partial Nephrectomy; Feasibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic Partial Nephrectomy (Active Comparator): Partial nephrectomy performed using the DaVinci robotic surgical system.
  Interventions: Procedure: Robotic Partial Nephrectomy
- Open Partial Nephrectomy (Active Comparator): Partial nephrectomy performed using the open approach.
  Interventions: Procedure: Open Partial Nephrectomy

INTERVENTIONS:
Procedure: Robotic Partial Nephrectomy — Robotic partial nephrectomy using da Vinci robot.
  Arms: Robotic Partial Nephrectomy
Procedure: Open Partial Nephrectomy — Standard open partial nephrectomy
  Arms: Open Partial Nephrectomy

SUMMARY:
A prospective randomized controlled feasibility trial for patients undergoing partial nephrectomy for T1 renal masses at Princess Margaret. Participants will be randomized receive either open or robotic partial nephrectomy.

DETAILED DESCRIPTION:
This is an interventional, unblinded RCT where a total of 30 patients who have consented to undergo partial nephrectomy for a T1 renal mass under the care of a uro-oncologist at Princess Margaret Cancer Centre will be randomized 1:1 to one of two arms:

Arm A: Robotic Partial Nephrectomy Arm B: Open Partial Nephrectomy

Patients will complete all pre-admission testing as per standard of care, regardless of arm allocation. Creatinine and eGFR are measured routinely pre-operatively and these values will be used as a baseline for all patients. In addition to standard pre-admission testing, participants will complete the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) offered either on paper at the visit or online via an emailed link.

Following either open or robotic partial nephrectomy, participants will be followed as per standard of care. Generally, this includes follow-up at 4-6 weeks, 6 months, 12 months and then either every 6 months thereafter or yearly, depending on pathology. All clinical outcome measures for this study are routinely reported post-operatively and in the follow-up period for partial nephrectomy patients. Quality of life will be assessed at the 4-7 week and 6 month follow-up visits using the EORTC QLQ-C30 offered either on paper at the visit or online via an emailed link. Participants will also be asked to complete a Surgical Recovery/Flank Bulge questionnaire regarding their incision healing and recovery from surgery at the 6-month follow-up visit.

The primary objective of this study is to assess the feasibility of a full RCT comparing perioperative outcomes in patients undergoing robotic vs. open partial nephrectomy at the investigator's institution.

The secondary objective of the study is to compare pilot outcome measures addressing oncologic, functional, and health economics outcomes to assess whether a full RCT is worthwhile and feasible.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically characterized T1 renal mass
* Elected for partial nephrectomy surgery
* Under the care of a uro-oncologist at Princess Margaret Cancer Centre
* Willing to comply with follow-up protocol
* Capable of providing informed consent

Exclusion Criteria:

* Radiologically characterized tumours ≥ T1
* Unfit for general anesthetic
* Unsuitable for robotic surgery (determined by treating physician)
* Unwilling to comply with standardized follow-up protocol
* Evidence of metastatic disease
* Solitary kidney
* Previous surgery on affected kidney
* Multiple tumours
* Known genetic syndromes predisposing to multiple renal tumours (e.g., VHL, TS, BHD)
* Pregnancy
* Inability to read, understand, and complete the questionnaires written in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-07-24 (Actual); Study Completion 2023-07-24 (Actual)

PRIMARY OUTCOMES:
Recruitment Potential | Study duration (2 years)
  Rate of accrual [participants per month]
Suitability of secondary outcome measures | Study duration (2 years)
  Assess the feasibility of collecting all secondary outcome data. To be assessed qualitatively by the study team and by calculating the proportion of patients with each data point completed.
Resource Utilization - Operating Room/Robotic Studio Time Availability | Study duration (2 years)
  Assess the capacity of accommodating surgical time for a full scale clinical trial. Measured by time from decision to treat to surgery date.
Resource Utilization - Cost of Study Participation | Study duration (2 years)
  To develop an accurate budget for a full trail, we are assessing the average cost of running the trial per patient, per arm. This calculation will include: cost of study coordinator time (number of hours x hourly wage), additional cost of robotic disposables, and cost of additional testing outside of standard of care.

SECONDARY OUTCOMES:
Operative Time | Duration of surgery
  Operative time in minutes
Warm Ischemia Time | Duration of surgery
  Measured in minutes from the time of application of first vascular clamp to removal of clamp
Blood Loss | Duration of surgery
  Estimated blood loss (mL), transfusion rates, use of hemostatic agents (which agents and how many used)
Conversion rate to radical nephrectomy or open partial nephrectomy | Duration of surgery
  Time in minutes from the start of robotic partial nephrectomy to the time decision was made to convert
Length of Stay | 1-7 days
  Calculated from day of admission to day of discharge
Complication Rates | Up to 6 months post-surgery
  Clavien-Dindo classification and need for/extent of re-intervention
Renal Function | Up to 6 months post-surgery
  Creatinine and eGFR measured pre-op, day 1 post-op, 4-7 weeks post-op, 6 months post-op
Positive margin rate | 1-3 weeks post-operatively
  Frequency of positive margins as reported in the final pathology report.
Margin size | 1-3 weeks post-operatively
  Distance from tumour to surgical margin (mm) as reported in final pathology report.
Analgesic Requirements | Up to 6 months post-operatively
  use of epidural, PCA, or oral analgesia
Quality of Life: EORTC QLQ-C30 | Up to 6 months post-operatively
  Measured using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) at 4-7 weeks and 6 months post-operatively
Surgical Recovery/Flank Bulge | 6 months from surgical date
  Surveyed at 6 months post-operatively
Health Economics | Study duration (2 years)
  Estimated overall cost of surgery for each arm (surgical supplies, length of stay, etc.) and cost of post-operative readmissions and ER visits

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada